CLINICAL TRIAL: NCT01147133
Title: Comparison of the Generic and Original Formulation of Clopidogrel Regarding the Potency of Platelet Inhibition in Patients After PCI
Brief Title: Comparison of Generic and Original Formulation of Clopidogrel
Acronym: DOSER-GENERIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pecs (Other)
Collaborators: Hungarian Academy of Sciences (Other); KRKA (Industry)
Responsible Party: Principal Investigator, Daniel Aradi MD, Assisstant Professor, University of Pecs
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: DOSER-GENERIC
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Heart Disease; Percutaneous Coronary Intervention
Keywords: Platelet aggregation; Generic; Clopidogrel; Comparison; VASP-PRI
MeSH Terms: conditions — Coronary Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Original (Experimental): Treatment phase with the original formulation of clopidogrel
  Interventions: Drug: Plavix
- Generic (Active Comparator): Treatment phase with the generic clopidogrel
  Interventions: Drug: Kardogrel

INTERVENTIONS:
Drug: Plavix — 1x75 mg
  Other Names: clopidogrel = PLAVIX
  Arms: Original
Drug: Kardogrel — 1x75 mg
  Other Names: generic clopidogrel = Kardogrel
  Arms: Generic

SUMMARY:
Clopidogrel is essential for the prevention of vascular events in patients after percutaneous coronary interventions (PCI). Most of our current knowledge with clopidogrel originates from the clinical investigations that had used Plavix®/Iscover® from Sanofi-Aventis as the original formulation of clopidogrel-bisulphate. However, as the patency of Plavix® has expired in November 2009 in Hungary, several generic clopidogrel have been introduced to the market. Some of the generics are using the original bisulphate formulation, while others are with besylate salt of clopidogrel. Despite the differences in the clopidogrel-salts, the different carriers might also modulate the pharmacokinetic/pharmacodynamic profile of each drug. As the consequences of the impaired antiplatelet potency might be devastating, including stent thrombosis, the investigators sought to compare generic clopidogrel to the original blister by different assays of platelet aggregation.

DETAILED DESCRIPTION:
Clopidogrel is essential for the prevention of vascular events in patients after percutaneous coronary interventions (PCI). Most of our current knowledge with clopidogrel originates from the clinical investigations that had used Plavix®/Iscover® from Sanofi-Aventis as the original formulation of clopidogrel-bisulphate. However, as the patency of Plavix® has expired in November 2009 in Hungary, several generic clopidogrel have been introduced to the market. Some of the generics are using the original bisulphate formulation, while others are with besylate salt of clopidogrel. Despite the differences in the clopidogrel-salts, the different carriers might also modulate the pharmacokinetic/pharmacodynamic profile of each drug. As the consequences of the impaired antiplatelet potency might be devastating, including stent thrombosis, the investigators sought to compare generic clopidogrel to the original blister by different assays of platelet aggregation.

In a prospective, cross-over, open-label, unblinded study the investigators aim to compare platelet activation and aggregation between Plavix® and generic clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the maintenance phase of PCI receiving 1x75 mg clopidogrel and 1x100 mg aspirin
* No planned interruption of the antiplatelet therapy in the next 1 month
* Informed consent

Exclusion Criteria:

* Oral anticoagulant therapy
* Contraindication for aspirin or clopidogrel
* Planned interruption of antiplatelet therapy in the next month

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
ADP 5 microM-induced maximal aggregation in light transmission aggregometry between the two time point. | 14 days

SECONDARY OUTCOMES:
VASP-PRI (%) 6-minute late aggregation with LTA (%) Proportion of patients with high platelet reactivity (HPR) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Aradi, MD PhD, Principal Investigator — University of Pécs, HUNGARY; András Komócsi, MD PhD, Study Director — University of Pécs, HUNGARY